CLINICAL TRIAL: NCT06130410
Title: COMIRNATY Intramuscular Injection for 6 Months to 4 Years Old (Monovalent: Omicron XBB.1.5) Special Investigation for Booster Immunization in Children Aged 6 Months to 4 Years
Brief Title: Special Investigation for Booster Dose of Comirnaty in Children Ages 6 Months Though 4 Years
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4591057
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: SARS-CoV-2; COVID-19
Keywords: COVID-19; SARS-CoV-2; Children (6 months though 4 years old); RNA Vaccine; Post-Marketing Study; Pediatric
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COMIRNATY intramuscular injection for 6 months to 4 years old (monovalent, omicron XBB.1.5.)
  Interventions: Biological: COMIRNATY intramuscular injection

INTERVENTIONS:
Biological: COMIRNATY intramuscular injection — Booster injection in the muscle, 1 dose

SUMMARY:
The purpose of this post-marketing study is to assess the safety of Comirnaty monovalent XBB.1.5. for booster vaccination children ages 6 months though 4 years under actual use medical practice.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 4 years at the time of the booster vaccination (4th dose) who (or whose representative) gave written consent to take part in the study.

Exclusion Criteria:

-There are no exclusion criteria for this study.

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children of 6 months though 4years of age, at the time of booster vaccination(4th dose)
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Local Country, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591057

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The enrollment period ended with 25 participants completed.
Groups:
- COMIRNATY Intramuscular Injection for 6 Months to 4 Years Old (Monovalent: Omicron XBB.1.5) 3μg: Participants aged 6 months to 4 years old were vaccinated with the booster (4th) dose of COMIRNATY intramuscular injection for 6 months to 4 years old (monovalent: Omicron XBB.1.5) on Day 1.
Period: Overall Study
Arm/Group | COMIRNATY Intramuscular Injection for 6 Months to 4 Years Old (Monovalent: Omicron XBB.1.5) 3μg
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A total of 25 participants were enrolled in this study. Of the 25 participants from whom case report forms (CRFs) were collected, no participants were excluded from the safety analysis set.
Arm/Group | COMIRNATY Intramuscular Injection for 6 Months to 4 Years Old (Monovalent: Omicron XBB.1.5) 3μg
Number analyzed (Participants) | 25
Age, Customized [Number; unit: participants]
  ≥6 months and <2 years | 15
  ≥2 and ≤4 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 13
  Sex: Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Adverse Reaction (AR)
Description: An adverse event was defined as any untoward medical occurrence attributed to COMIRNATY intramuscular injection for 6 months to 4 years old (monovalent: Omicron XBB.1.5) in a participant who was vaccinated. The relatedness was assessed by the physician. Events for which a causal relationship with intramuscular injection could not be ruled out were handled as ARs.
Time Frame: For 28 days after the booster (4th) dose
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and were vaccinated with COMIRNATY intramuscular injection for 6 months to 4 years old (monovalent: Omicron XBB.1.5) at least once. Among the 25 participants with fixed CRFs in the study, no participants were excluded from the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | COMIRNATY Intramuscular Injection for 6 Months to 4 Years Old (Monovalent: Omicron XBB.1.5) 3μg
Number analyzed (Participants) | 25
Participants | 1

2. Primary Outcome: Proportion of Participants With Serious Adverse Reaction (SAR)
Description: An SAR was defined as any AR resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening; hospitalization or prolongation of existing hospitalization; persistent or significant disability/malfunction; congenital anomaly/birth defect; or other medically important events.
Time Frame: For 28 days after the booster (4th) dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | COMIRNATY Intramuscular Injection for 6 Months to 4 Years Old (Monovalent: Omicron XBB.1.5) 3μg
Number analyzed (Participants) | 25
Participants | 0

3. Primary Outcome: Proportion of Participants With Reactogenicity (≥ Grade 1) in Those Who Are Younger Than 2 Years of Age
Description: Local reactions and systemic events recorded in the health observation diary collected by the physician from study participants were handled as reactogenicity events.
  They were aggregated for the vaccinated participants by age group and grade. The results were aggregated by age group for local reactions and systemic events of grade 1 or higher.
  If the participants were younger than 2 years of age on the date of the booster (4th) dose, the following reactogenicity events were aggregated. Local reactions: injection site tenderness, redness, and injection site swelling. Systemic events: pyrexia, decreased appetite, somnolence, and irritability. If the participants were 2 years or older on the date of the booster (4th) dose, the following reactogenicity events were aggregated. Local reactions: injection site pain, redness, and injection site swelling. Systemic events: pyrexia, vomiting, diarrhoea, headache, malaise, chills, myalgia, and arthralgia.
Time Frame: Within 7 days after the date of the booster (4th) dose
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and were vaccinated with COMIRNATY intramuscular injection for 6 months to 4 years old (monovalent: Omicron XBB.1.5) at least once. Among the 25 participants with fixed CRFs in the study, no participants were excluded from the safety analysis set. Of the safety analysis set, participants younger than 2 years were included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Participants Younger Than 2 Years of Age Who Were Vaccinated With COMIRNATY Intramuscular Injection: Participants younger than 2 years were vaccinated with the booster (4th) dose of COMIRNATY intramuscular injection for 6 months to 4 years old (monovalent: Omicron XBB.1.5).
Arm/Group | Participants Younger Than 2 Years of Age Who Were Vaccinated With COMIRNATY Intramuscular Injection
Number analyzed (Participants) | 15
Participants
  Local reactions (Grade 1 or higher) | 5
  Systemic events (Grade 1 or higher) | 4

4. Primary Outcome: Proportion of Participants With Reactogenicity (≥ Grade 1) in Those Who Are Aged 2 Years or Older
Description: as for outcome 3
Time Frame: Within 7 days after the date of the booster (4th) dose
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and were vaccinated with COMIRNATY intramuscular injection for 6 months to 4 years old (monovalent: Omicron XBB.1.5) at least once. Among the 25 participants with fixed CRFs in the study, no participants were excluded from the safety analysis set. Of the safety analysis set, participants aged 2 years or older were included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Participants Aged 2 Years or Older Who Were Vaccinated With COMIRNATY Intramuscular Injection: Participants aged 2 years or older were vaccinated with the booster (4th) dose of COMIRNATY intramuscular injection for 6 months to 4 years old (monovalent: Omicron XBB.1.5).
Arm/Group | Participants Aged 2 Years or Older Who Were Vaccinated With COMIRNATY Intramuscular Injection
Number analyzed (Participants) | 10
Participants
  Local reactions (Grade 1 or higher) | 7
  Systemic events (Grade 1 or higher) | 2

ADVERSE EVENTS:
Time Frame: For 28 days after the booster (4th) dose
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | COMIRNATY Intramuscular Injection for 6 Months to 4 Years Old (Monovalent: Omicron XBB.1.5) 3μg
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 5/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | COMIRNATY Intramuscular Injection for 6 Months to 4 Years Old (Monovalent: Omicron XBB.1.5) 3μg (N=25)
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT06130410/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-24): https://cdn.clinicaltrials.gov/large-docs/10/NCT06130410/SAP_001.pdf